CLINICAL TRIAL: NCT04113135
Title: The Utilization of Yoga as a Therapeutic Tool to Promote Physical Activity Behavior Change and Improved Postural Control in Individuals With Multiple Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete initial data collection due to tornado and then COVID-19 has limited in person data collection/intervention.
Sponsor: Winston Salem State University (Other)
Collaborators: Appalachian State University (Other)
Responsible Party: Principal Investigator, LaVerene M Garner, PT, DPT; Visiting Clinical Assistant Professor;, Winston Salem State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0118
Record Dates: First submitted 2019-08-29; First posted 2019-10-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers and participants will not be blinded due to the nature of the intervention. Participants will know whether or not they are performing yoga or just receiving the control group intervention. Additionally, the PI is leading the intervention and will therefore know who is in the control vs the experimental. Investigators will attempt to blind clinicians and students completing pre and post intervention testing to who was in the control vs experimental, however, this may not be possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Journaling, meditations, education, yoga intervention Arm (Experimental): Participants will be required to attend 1x/wk for 7 total sessions. The pre/post testing will take approximately 45 minutes to one hour. Session 1 for all participants will be comprised of an initial screening with a health history questionnaire regarding information about comorbidities, medications, and type of Multiple Sclerosis (MS) diagnosis, and completion of all outcome measurement tests as listed above. Following session one, subjects will be assigned to the control or experimental group utilizing the robust randomization application (RRApp) and the block randomization technique to ensure an equal number of subjects in each group.39 The intervention sessions (2-6) for the experimental group participants consist will include a group discussion of the objectives for the week, 20-30 minutes of education and journaling (Attachment B), 45-60 minutes of PA consisting of various yoga poses followed by SMART goal setting and guided relaxation..
  Interventions: Other: Yoga
- Journaling, meditation, education arm (Active Comparator): Participants will be required to attend 1x/wk for 7 total sessions. The pre/post-testing will take approximately 45 minutes to one hour. Session 1 for all participants (control and experimental) will be comprised of an initial screening with a health history questionnaire regarding information about comorbidities, medications, and type of Multiple Sclerosis (MS) diagnosis, and completion of all outcome measurement tests as listed above. Following session one, subjects will be assigned to the control or experimental group utilizing the robust randomization application (RRApp) and the block randomization technique to ensure an equal number of subjects in each group.39 The control group will participate in a 45-60 minute session for weeks 2-6 consisting of goal setting to facilitate behavior change, education on MS, and meditation. Session 7 will conclude the study with reassessment of all outcome measurements as listed above.
  Interventions: Other: Control

INTERVENTIONS:
Other: Yoga — Participants will be lead through a series of yoga poses by a licensed physical therapist with advanced training in yoga. Participants in this group will also receive education related to MS as well as SMART goal setting, journaling and guided meditation. Modifications will be offered as needed.
  Arms: Journaling, meditations, education, yoga intervention Arm
Other: Control — Participants in this group will receive education related to MS as well as SMART goal setting, journaling, and guided meditation.
  Arms: Journaling, meditation, education arm

SUMMARY:
This randomized control trial will investigate whether using yoga as physical activity improves quality of life, self-efficacy for physical activity, reactive balance, and dual tasking more than education, journaling, and meditation alone in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune disease characterized by chronic inflammation specifically targeting the central nervous system. 1 It is associated with destruction of the surrounding myelin sheaths leading to formation of plaques/lesions dispersed throughout the brain and spinal cord. 1 The prevalence of MS is nearly one million in the United States with the majority of diagnoses occurring between the ages of 20 and 50. 2 Though the precise etiology remains unknown, genetic and environmental factors have been linked to the cause and therefore MS is considered a multifactorial disease. 3 Hallmark signs of MS include progressive demyelination, oligodendrocyte damage, and ultimately axonal destruction. These adaptations occur due to an inflammatory response consisting of macrophages, microglia, T and B Cells, followed by an intense astrocyte reaction leading to glial scarring, a common characteristic of chronic MS lesions. 4 According to Lassmann 1, clinical deficits seen throughout the course of MS are more closely correlated to the degree of axonal loss as opposed to the amount of lesions or extent of demyelination. These include deficits in cognition, vision, bowel and bladder control, coordination, and loss of muscle strength. 5 Multiple Sclerosis has various subtypes making the clinical course heterogeneous among patients. 6 Subtypes include: clinically isolated syndrome (CIS), relapsing remitting MS (RRMS), primary progressive MS (PPMS), and secondary progressive MS (SPMS). 6 The variability of disease course for each individual subtype is extremely important, and should be taken into consideration for prognosis and intervention options. 3

Due to the aggressive, progressive, unpredictable nature of MS, lack of evidence for a cure, and the wide array of cognitive and physical symptoms, MS can detrimentally impact a patient's health and reduce overall quality of life. 7 Current research advocates for physical activity (PA) as an intervention to combat these effects. Physical activity is referred to here as low to moderate level exercise. 8 Some individuals with MS who incorporated long-term physical activity into their life demonstrated a decrease in the progression of the disease and a reduction in MS flare-ups. 9 In order to successfully implement PA based interventions for the management of MS one must first identify individual motivators for PA. 5 Motivators for physical activity include self-efficacy and internalized motivation which are derived from physical activity outcomes. 5Self-efficacy is "the belief that one can successfully cope with challenging conditions" 7 whereas self -determination refers to the origin of one's motivation. 8 Other researchers found that "those with MS who were more physically active had greater self-efficacy for function and control, and self-efficacy for function and control were associated with greater physical and psychological components of quality of life." 7 However, the vast majority of those diagnosed with MS avoid exerting themselves due to symptoms of muscle weakness and fatigue; this lack of PA is thought to exacerbate those symptoms which then leads to a perpetual cycle of inactivity and flare-ups. 8,9 Therefore, it has also been theorized that a program designed for MS patients which focuses on promoting self-efficacy could lead to long-term PA participation and thus result in increased quality of life. 8

One such form of physical activity that could provide physiological and psychological benefits for individuals diagnosed with MS is yoga. "Yoga is an ancient Indian, non-religious mind- body approach that has components centering on meditation, mindfulness, breathing, and activity or postures." 10 Exercise programs which involve these components have been found to improve the quality of life by addressing the biopsychosocial (BPS) model. The BPS model is composed of biological, psychological and social components which has been found to have a positive impact on an individual's health. 11 Therefore, it is hypothesized that by increasing muscular strength and flexibility while decreasing affective factors such as depression, stress and anxiety and improving social factors will improve an individual's overall well-being and allow them to cope with the symptoms associated with MS. 11,12 Numerous studies have found yoga to be beneficial in improving fatigue and other symptoms associated with MS. 13 For example, standing yoga poses can promote improved reactive balance through the use of stepping strategies. Yoga also has the potential to reduce cognitive and motor costs for individuals during dual tasks resulting in decreased interference and thus optimal functioning in more challenging conditions. 14 Previous research has demonstrated that yoga significantly improved "physical performance and mental function" and factors associated with quality of life in subjects with MS.15 Based on these findings, the investigators hypothesize that yoga will improve quality of life and self-efficacy for physical activity in people living with MS.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Multiple Sclerosis.

PDDS Category 0-6. Those patients that are classified as PDDS 5 or 6, must be able to ambulate into the clinic without the use of a wheelchair or scooter.

Ability to participate in light to moderate physical activity for 45 minutes one time per week.

-

Exclusion Criteria:

Participants experiencing a multiple sclerosis exacerbation at the time of the scheduled intervention

Serious Cardiovascular Disease (Uncompensated CHF, Unmanaged hypertension)

Advanced Musculoskeletal Disorder (ie. Unhealed Fracture, advanced stages of osteoporosis)

PDDS Category 7-8

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini BESTest (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  Participants will each complete the Mini Balance Evaluation Systems Test (MiniBEST).
  This assessment is a series of 14 tests measuring anticipatory balance, reactive postural control, sensory orientation, and dynamic gait. 16 The 14 tests will be analyzed together to determine reactive and anticipatory balance, as well as, dual task capabilities. Subjects will be tested with flat-heeled shoes or with shoes and socks off. 16 Each of the 14 items are scored on an ordinal scale from 0-2 with a total of 28 points possible. Higher scores indicate higher levels of function, with 0 indicating the lowest level of function and 2 indicating the highest level of function. Two of the 14 items (Item 3 and Item 6) have right and left assessments in which the lower of the two sides is calculated into the total. If an assistive device is used during an item the score is lowered by one point. If the participant requires physical assistance then the item is automatically scored a 0. 16
9 hole peg test (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  Test of fine motor coordination where subjects are asked to use their hands to move 9 pegs from one side of a tray to another. This is a timed outcome.
Timed 25 ft walk (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  Subjects are asked to walk 25 ft over level surfaces and are timed
Markus Self-Efficacy Scale (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  The Marcus Self Efficacy Scale is a survey which will be used to measure participants' beliefs about their ability to exercise. 23 This scale consists of five items that resemble barriers to exercise such as planning time, environmental factors, and physical or emotional well-being. 23 For each scenario, participants rate their confidence on an 11-point Likert scale; 0 is 'does not apply to me,' 1 is 'not at all confident' and 11 is 'very confident.' 23 Lower scores indicate lower self-efficacy and suggest less inclination to participate in exercise. According to Marcus et al, this scale scored a test-retest reliability of r=.90 over a two-week period.
Quality of Life Scale (Change is being assessed) | Pre and post intervention(Week 1 of protocol and week 7 of protocol)
  The Quality of Life (QoL) survey consists of 32 items created by Gill et al. 24 This survey allows the participant to evaluate their quality of life based on the biopsychosocial model. The participants are asked to circle a number from 1 'poor' to 5 'excellent' based on their perception of their quality of life. Gill et al 24 recommended the QoL survey as a valuable tool in research based on its psychometric properties. Gill et al 25 re-evaluated the QoL survey for test-retest reliability and compared to other quality of life measurements. Gill et al 24 reported reliability of .793 for ADL and .950 for spirituality. In addition, the QoL survey demonstrated good test-retest reliability ranging from .677 to .816, and intraclass correlations from .676 to .809. 25
Patient Determined Disease Steps (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  The Patient Determined Disease Steps (PDDS) will be completed by participants in order to determine their level of disability based on their method of ambulation. 26 This outcome measure is based on the Disease Steps scale created by Hohol et al 27 which sought to provide neurologists with a simple guide for therapeutic intervention and to assess patient progress. The PDDS consists of nine ordinal rankings from 0 (normal) to 8 (bedridden). The PDDS has a strong correlation with the Expanded Disability Status Scale (EDSS) which is the most widely accepted measure for MS disability; this confirms criterion validity. 26 According to Learmonth et al 26 the PDDS is a valid and useful patient-reported score system for assessing disability in individuals with MS.
Modified Fatigue Impact Scale (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  The Modified Fatigue Impact Scale (MFIS) is a self-reported survey which will be used to determine the impact of fatigue on an individual over the last four weeks. 28 This consists of twenty-one items rated on a 5-point Likert scale with 0 being 'never' and 4 being 'almost always'. Scores can be subdivided into physical, psychosocial, and cognitive subscales. Total scores range from 0-84 with higher scores indicating greater fatigue and MS related fatigue is identified as a score of 38 or greater. 28 The minimal clinically important change for the MFIS is 16 points short-term and 20 points long-term. 28 Learmonth et al 28 found the MFIS has an excellent test-retest reliability of 0.837 over a 6-month period. In addition, Amtmann et al 29 found that the MFIS has excellent internal consistency, demonstrated by a Cronbach's alpha greater than 0.93, and known groups validity.
Pittsburgh Sleep Quality Index (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  The Pittsburgh Sleep Quality Index (PSQI) is a 19 item self-rated questionnaire that will be completed by the participants. The PSQI will serve as a subjective measure of sleep for participants participating in the study, and allow for discrimination between "good" and "poor" sleepers. 30 The 19 individual items assessed help to generate seven component, consisting of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. 30 A global score is obtained from the seven components, ranging from 0-21, with higher scores reflecting poor sleep quality. 31 While the PSQI has not been specifically validated in people diagnosed with MS, it has been used to assess changes in sleep patterns in those diagnosed with MS in many different studies. 30,31
Godin Leisure-Time Physical Activity Questionnaire (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  The Godin is a 3-question, self-report measure that assesses the frequency that individuals engage in bouts of PA at light, moderate, and strenuous levels. 34 The measure asks frequency of PA at each activity level and uses a formula to calculate a score (MET value) for weekly activity (9 x strenuous, 5 x moderate, and 3 x light). The higher the overall score, the greater the PA level. The MET scores can also be used to classify PA participation into three categories: "active" (24 and higher), "moderately active" (14-23), and "insufficiently active" (less than 14). More recently, research has proposed using only using the moderate and strenuous calculations to classify individuals as "active" (? 24 METS) and insufficiently active" (? 23 METS) to fall in line with PA guidelines in both the United States and Canada. 35-36 It has been used extensively with the MS population. 38
Basic Demographics and Behavioral questionnaire (Change is being assessed) | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  A basic background questionnaire will be used to gather information on participants age, gender, work history, history with MS, and leisure and physical activity behavior.
Bladder control scale | Pre and post intervention (Week 1 of protocol and week 7 of protocol)
  The Bladder Control Scale (BLCS) is a survey consisting of four items that briefly assess bladder. control and the impact it has on the individual's quality of life. This survey was developed by Turnbull et al (1992) and is cited by the National Multiple Sclerosis user's manual and Beadnall et al. 32 The BLCS has a scoring system ranging from 0-22 with higher scores indicating more difficulty with bladder control. 32, 33 MS specialists were consulted during the development of this scale to ensure content validity. Beadnall et al 32 noted multiple studies showing the BLCS to be valid and having good reliability.

CONTACTS AND LOCATIONS:
Overall Officials: LaVerene Garner, DPT, Principal Investigator — Winston Salem State University
Locations (1):
- Winston Salem State University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be de-identified using a number system to ensure the privacy of the individual's health data. Hard copy data will be double-locked in a secure location at Winston Salem State University. Electronic data will be stored on a password protected computer. Data collected will only be accessible to the principal and supplementary investigators. Data will be saved for a minimum of three years. Individuals who will have access to de-identified data will include the principal investigator, co-investigators (Dr Fasczewski and Dr Migliarese), and student physical therapists who are functioning in a graduate assistant role during the study. Additionally, we plan to submit for a clinical trial registry number. No other individuals will have access to individual data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available as collected and will be available through the conclusion of the study (potentially two years)
Access Criteria: CITI training and IRB approval

REFERENCES:
- [Background] Lassmann H. Neuropathology in multiple sclerosis: new concepts. Mult Scler. 1998 Jun;4(3):93-8. doi: 10.1177/135245859800400301. PMID 9762654
- [Background] National Multiple Sclerosis Society. Who Gets MS? (Epidemiology). https://www.nationalmssociety.org/What-is-MS/Who-Gets-MS. Accessed June 9, 2019
- [Background] Ghasemi N, Razavi S, Nikzad E. Multiple Sclerosis: Pathogenesis, Symptoms, Diagnoses and Cell-Based Therapy. Cell J. 2017 Apr-Jun;19(1):1-10. doi: 10.22074/cellj.2016.4867. Epub 2016 Dec 21. PMID 28367411
- [Background] Bruck W, Lucchinetti C, Lassmann H. The pathology of primary progressive multiple sclerosis. Mult Scler. 2002 Apr;8(2):93-7. doi: 10.1191/1352458502ms785rr. PMID 11990878
- [Background] Fasczewski KS, Rothberger SM, Gill DL. Why do they do it? Assessing self-report physical activity behavior and quality of life in individuals with multiple sclerosis. J Health Psychol. 2020 Jun;25(7):964-975. doi: 10.1177/1359105317739965. Epub 2017 Nov 27. PMID 29172811
- [Background] Hurwitz BJ. The diagnosis of multiple sclerosis and the clinical subtypes. Ann Indian Acad Neurol. 2009 Oct;12(4):226-30. doi: 10.4103/0972-2327.58276. PMID 20182569
- [Background] Motl RW, Snook EM. Physical activity, self-efficacy, and quality of life in multiple sclerosis. Ann Behav Med. 2008 Feb;35(1):111-5. doi: 10.1007/s12160-007-9006-7. Epub 2008 Feb 12. PMID 18347911
- [Background] Fasczewski KS, Gill DL. A model of motivation for physical activity in individuals diagnosed with multiple sclerosis. Disabil Rehabil. 2019 Sep;41(18):2143-2150. doi: 10.1080/09638288.2018.1459883. Epub 2018 Apr 10. PMID 29631465
- [Background] Fasczewski KS, Gill DL, Rothberger SM. Physical activity motivation and benefits in people with multiple sclerosis. Disabil Rehabil. 2018 Jun;40(13):1517-1523. doi: 10.1080/09638288.2017.1300946. Epub 2017 Mar 14. PMID 28291956
- [Background] Wahbeh H, Elsas SM, Oken BS. Mind-body interventions: applications in neurology. Neurology. 2008 Jun 10;70(24):2321-8. doi: 10.1212/01.wnl.0000314667.16386.5e. PMID 18541886
- [Background] Bolton RE, Fix GM, VanDeusen Lukas C, Elwy AR, Bokhour BG. Biopsychosocial benefits of movement-based complementary and integrative health therapies for patients with chronic conditions. Chronic Illn. 2020 Mar;16(1):41-54. doi: 10.1177/1742395318782377. Epub 2018 Jun 18. No abstract available. PMID 29914264
- [Background] Kahraman T, Ozdogar AT, Yigit P, Hosgel I, Mehdiyev Z, Ertekin O, Ozakbas S. Feasibility of a 6-Month Yoga Program to Improve the Physical and Psychosocial Status of Persons with Multiple Sclerosis and their Family Members. Explore (NY). 2018 Jan-Feb;14(1):36-43. doi: 10.1016/j.explore.2017.07.006. Epub 2017 Oct 23. PMID 29174060
- [Background] Rogers KA, MacDonald M. Therapeutic Yoga: Symptom Management for Multiple Sclerosis. J Altern Complement Med. 2015 Nov;21(11):655-9. doi: 10.1089/acm.2015.0015. Epub 2015 Aug 13. PMID 26270955
- [Background] Subramaniam S, Bhatt T. Effect of Yoga practice on reducing cognitive-motor interference for improving dynamic balance control in healthy adults. Complement Ther Med. 2017 Feb;30:30-35. doi: 10.1016/j.ctim.2016.10.012. Epub 2016 Oct 26. PMID 28137524
- [Background] Cohen ET, Kietrys D, Fogerite SG, Silva M, Logan K, Barone DA, Parrott JS. Feasibility and Impact of an 8-Week Integrative Yoga Program in People with Moderate Multiple Sclerosis-Related Disability: A Pilot Study. Int J MS Care. 2017 Jan-Feb;19(1):30-39. doi: 10.7224/1537-2073.2015-046. PMID 28243184
- [Background] King L, Horak F. On the mini-BESTest: scoring and the reporting of total scores. Phys Ther. 2013 Apr;93(4):571-5. doi: 10.2522/ptj.2013.93.4.571. No abstract available. PMID 23547173
- [Background] Ross E, Purtill H, Uszynski M, Hayes S, Casey B, Browne C, Coote S. Cohort Study Comparing the Berg Balance Scale and the Mini-BESTest in People Who Have Multiple Sclerosis and Are Ambulatory. Phys Ther. 2016 Sep;96(9):1448-55. doi: 10.2522/ptj.20150416. Epub 2016 Feb 25. PMID 26916925
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Feys P, Lamers I, Francis G, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. The Nine-Hole Peg Test as a manual dexterity performance measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):711-720. doi: 10.1177/1352458517690824. Epub 2017 Feb 16. PMID 28206826
- [Background] Yozbatiran N, Baskurt F, Baskurt Z, Ozakbas S, Idiman E. Motor assessment of upper extremity function and its relation with fatigue, cognitive function and quality of life in multiple sclerosis patients. J Neurol Sci. 2006 Jul 15;246(1-2):117-22. doi: 10.1016/j.jns.2006.02.018. Epub 2006 May 5. PMID 16678208
- [Background] Fischer JS, Rudick RA, Cutter GR, Reingold SC. The Multiple Sclerosis Functional Composite Measure (MSFC): an integrated approach to MS clinical outcome assessment. National MS Society Clinical Outcomes Assessment Task Force. Mult Scler. 1999 Aug;5(4):244-50. doi: 10.1177/135245859900500409. PMID 10467383
- [Background] Motl RW, Cohen JA, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the timed 25-foot walk as an ambulatory performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):704-710. doi: 10.1177/1352458517690823. Epub 2017 Feb 16. PMID 28206828
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Gill DL, Chang Y, Murphy KM et al. Quality of Life Assessment for Physical Activity and Health Promotion. Applied Research in Quality of Life. 2011 June; 6(2):181-200
- [Background] Gill DL, Reifsteck EJ, Adams MM, Shang Y. Quality of Life Assessment for Physical Activity and Health Promotion: Further Psychometrics and Comparison of Measures. Measurement in Physical Education & Exercise Science 2015 Oct;19(4):159-166.
- [Background] Learmonth YC, Motl RW, Sandroff BM, Pula JH, Cadavid D. Validation of patient determined disease steps (PDDS) scale scores in persons with multiple sclerosis. BMC Neurol. 2013 Apr 25;13:37. doi: 10.1186/1471-2377-13-37. PMID 23617555
- [Background] Hohol MJ, Orav EJ, Weiner HL. Disease steps in multiple sclerosis: a simple approach to evaluate disease progression. Neurology. 1995 Feb;45(2):251-5. doi: 10.1212/wnl.45.2.251. PMID 7854521
- [Background] Learmonth YC, Dlugonski D, Pilutti LA, Sandroff BM, Klaren R, Motl RW. Psychometric properties of the Fatigue Severity Scale and the Modified Fatigue Impact Scale. J Neurol Sci. 2013 Aug 15;331(1-2):102-7. doi: 10.1016/j.jns.2013.05.023. Epub 2013 Jun 20. PMID 23791482
- [Background] Amtmann D, Bamer AM, Noonan V, Lang N, Kim J, Cook KF. Comparison of the psychometric properties of two fatigue scales in multiple sclerosis. Rehabil Psychol. 2012 May;57(2):159-66. doi: 10.1037/a0027890. PMID 22686554
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Trojan DA, Arnold D, Collet JP, Shapiro S, Bar-Or A, Robinson A, Le Cruguel JP, Ducruet T, Narayanan S, Arcelin K, Wong AN, Tartaglia MC, Lapierre Y, Caramanos Z, Da Costa D. Fatigue in multiple sclerosis: association with disease-related, behavioural and psychosocial factors. Mult Scler. 2007 Sep;13(8):985-95. doi: 10.1177/1352458507077175. Epub 2007 Apr 27. PMID 17468448
- [Background] Beadnall HN, Kuppanda KE, O'Connell A, Hardy TA, Reddel SW, Barnett MH. Tablet-based screening improves continence management in multiple sclerosis. Ann Clin Transl Neurol. 2015 Jun;2(6):679-87. doi: 10.1002/acn3.205. Epub 2015 May 1. PMID 26125042
- [Background] Ritvo P, Fischer J, Miller D, et al. Multiple sclerosis quality of life inventory: a user's manual. National Multiple Sclerosis Society: New York, United States of America, 1997. p. 1-35.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Amireault S, Godin G. The Godin-Shephard leisure-time physical activity questionnaire: validity evidence supporting its use for classifying healthy adults into active and insufficiently active categories. Percept Mot Skills. 2015 Apr;120(2):604-22. doi: 10.2466/03.27.PMS.120v19x7. Epub 2015 Mar 23. PMID 25799030
- [Background] Godin G. The Godin-Shephard Leisure-Time Physical Activity Questionnaire. Health Fit J Cananda. 2011;4(1):18-22.
- [Background] Jacobs DR Jr, Ainsworth BE, Hartman TJ, Leon AS. A simultaneous evaluation of 10 commonly used physical activity questionnaires. Med Sci Sports Exerc. 1993 Jan;25(1):81-91. doi: 10.1249/00005768-199301000-00012. PMID 8423759
- [Background] Motl RW, McAuley E. Physical activity and health-related quality of life over time in adults with multiple sclerosis. Rehabil Psychol. 2014 Nov;59(4):415-421. doi: 10.1037/a0037739. Epub 2014 Aug 25. PMID 25150806
- [Background] Tu C, Benn EKT. RRApp, a robust randomization app, for clinical and translational research. J Clin Transl Sci. 2017 Dec;1(6):323-327. doi: 10.1017/cts.2017.310. Epub 2018 Feb 19. PMID 29707253